CLINICAL TRIAL: NCT06105437
Title: BE-EMPOWERed Study: Belgian Study Enhancing the Uptake and the Effectiveness of a Multifactorial Falls Prevention Intervention in Older Community-dWElling peRsons
Brief Title: Implementation of a Multifactorial Falls Prevention Intervention in Older Community-dWElling peRsons
Acronym: BE-EMPOWERed
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: KU Leuven (Other)
Collaborators: Flemish Agency for Care and Health (Other)
Responsible Party: Principal Investigator, prof. dr. Koen Milisen, Prof. dr., KU Leuven
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: BE-EMPOWERed
Record Dates: First submitted 2023-10-12; First posted 2023-10-27 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Falls Prevention; Implementation; Older People
Keywords: Community setting; Implementation; Falls prevention; Aged

STUDY DESIGN:
Intervention Model Description: A mixed methods study with a convergent parallel design will be carried out in four primary care areas in Flanders (Belgium). Within this mixed methods study, the researchers gather information on and experiences with the implementation process of the BE-EMPOWERed program from the perspective of the older people, healthcare professionals, implementation facilitators, the working group of the primary care area and local policy makers. To evaluate the implementation process and outcomes, the following data are being collected: reach, fidelity, feasibility, acceptability, sustainability and cost of implementation. A variety of methods are being used to collect data on implementation outcomes and process such as self-reported implementation costs, surveys, interviews and focus groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BE-EMPOWERed program (Other): The BE-EMPOWERed program entails a group program for older people, workshops for healthcare professionals and a 6-steps implementation plan for primary care areas. The group program for older people is based on the main principles of the Australian multifactorial falls prevention program 'Stepping On'. The workshops for healthcare professionals focus on the multifactorial falls prevention approach, reimbursement of healthcare costs, referrals to other healthcare professionals and motivational interviewing. The Implementation plan consists of 6-steps: 1. enable support, 2. map baseline situation, 3. define objectives and priorities, 4. plan implementation, 5. implementation and 6. evaluation, adjust and work towards sustainability. Last, to support the primary care areas, implementation facilitators were trained.
  Interventions: Other: BE-EMPOWERed program

INTERVENTIONS:
Other: BE-EMPOWERed program — The BE-EMPOWERed program entails a group program for older people, workshops for healthcare professionals and a 6-steps implementation plan for primary care areas. The group program for older people is based on the main principles of the Australian multifactorial falls prevention program 'Stepping On'. The workshops for healthcare professionals focus on the multifactorial falls prevention approach, reimbursement of healthcare costs, referrals to other healthcare professionals and motivational interviewing. The Implementation plan consists of 6-steps: 1. enable support, 2. map baseline situation, 3. define objectives and priorities, 4. plan implementation, 5. implementation and 6. evaluation, adjust and work towards sustainability. Last, to support the primary care areas, implementation facilitators were trained.

SUMMARY:
Approximately 24 to 40% community-dwelling older persons fall annually, of which 21 to 45% fall recurrently. Many factors contribute to the risk of falling, such as mobility impairment, medication use, environmental issues and risk behavior. Falls are associated with an increased risk of morbidity and mortality and often lead to physical and psychosocial consequences. Falls and related injuries have a huge economic impact on society. Given its proven efficacy as shown by controlled trials, multifactorial falls prevention interventions are recommended as primary strategy. However, poor implementation in daily clinical practice leads to inconclusive results on clinical outcomes. Several studies show that implementation, effectiveness and context are linked. Context is a critical concept to understand variation in implementation and clinical outcomes. Therefore, it is necessary to comprehensively understand the context prior to implementation.To date, the context and tailored implementation are neglected in the majority of falls prevention research. Given this, this Belgian study aims to Enhance the uptake and the Effectiveness of a Multifactorial falls Prevention intervention in Older community-dWElling peRsons (BE-EMPOWERed).

DETAILED DESCRIPTION:
The overall objective is to comprehensively evaluate the BE-EMPOWERed program on clinical and implementation outcomes and assess the implementation processes.The BE-EMPOWERed program consists of a multifactorial falls prevention intervention in older persons and strategies to implement the intervention, both tailored to the community setting in Belgium (Flanders).

Aim: To implement the BE-EMPOWERed program in 4 primary care areas in Belgium (Flanders) and to explore the effectiveness on clinical outcomes and to assess the implementation process and outcomes in a mixed methods study with a convergent parallel design.

i. To explore the effectiveness of the BE-EMPOWERed program on fear of falling.

ii. To assess the implementation outcomes for the BE-EMPOWERed program such as: reach, fidelity, feasibility, acceptability, sustainability and implementation costs.

iii. To understand the implementation process of the BE-EMPOWERed program from the perspective of the older persons, healthcare professionals, local service centers and local policy makers.

Overall methodology: We use Intervention Mapping in line with the Medical Research Council (MRC) framework for developing and evaluating the BE-EMPOWERed program.

A stakeholder group is installed and meets twice each year during the development, implementation and evaluation (October 2020 - December 2025). It includes 21 participants: two physiotherapists, an occupational therapist, a geriatrician and a pharmacist; a representative of the local service centers in Flanders, of the Flemish council of older persons and of Flanders Institute of Healthy Living and two representatives of 'Lokaal Gezondheids Overleg' (LOGO); a researcher in occupational therapy; a researcher in physiotherapy and a researcher with expertise in implementation science; a staff member of a home care nursing organization, of an organization of home health aides, of an organization that represents family caregivers and home care districts in Flanders, of an organization that represents general practitioners, of a Belgian sickness funds and of the Center of Expertise for Falls and Fracture Prevention Flanders; a policy maker of the Flemish Government and a coach for older persons.

Setting: Flanders has 6.7 million inhabitants, has five provinces and consists of 59 primary care areas. A primary care area is developed by the Flemish Government and is network of primary care providers in a geographically defined area; with the objective to exchange knowledge and information and to coordinate their activities. The study takes place in 4 primary care areas.

Evaluation: A mixed methods study with a convergent parallel design in 4 primary care areas. A variety of methods are being used to collect data on implementation outcomes and process such as self-reported implementation costs, surveys, interviews and focus groups.

ELIGIBILITY:
Inclusion Criteria group program:

* Community-dwelling
* 65 years and over
* Independent with or without walking aid
* Understanding and speaking of the Dutch language
* Experienced one or more of the following events in the past year? (1) one or more falls; or (2) mobility or balance problems; or (3) concerns about falling

Exclusion Criteria group program:

- Neurological and cognitive problems (Parkinson, CVA, dementia, delirium)

Inclusion Criteria workshops:

* Healthcare professionals
* Working in the primary care area
* Understanding and speaking of the Dutch language

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 550 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Fidelity of the group program | Immediately after every session and follow-up session (up to 8 months).
  Fidelity is defined as the degree to which an intervention was implemented as it was prescribed in the original protocol or as it was intended by the program developers.
  Based on the key elements of the group program a questionnaire was developed (fidelity checklist). After every group program the group leader will fill in this questionnaire. The researcher will also observe one out of seven sessions and give feedback to the group leader based on the key elements of this questionnaire (fidelity checklist).
  The percentage of key elements that were complied or not complied to by the group leader will be measured.
Fidelity of the workshops | Immediately after every workshop (up to 1 month).
  Fidelity is defined as the degree to which an intervention was implemented as it was prescribed in the original protocol or as it was intended by the program developers.
  Fidelity checklist by the trainer. Based on the key elements of the workshops a questionnaire was developed (fidelity checklist). After every workshop the trainer will fill in this questionnaire (self reporting) The percentage of key elements that were complied or not complied to by the trainer will be measured.

SECONDARY OUTCOMES:
Reach older people | Immediately after every session and follow-up session (up to 8 months).
  Reach is defined as the absolute number, proportion, and representativeness of individuals who are willing to participate in a given initiative, intervention, or program, and reasons why or why not.
  Reach of the older people. Participant list group program by the group leader.
Implementation cost | 2 years
  Is defined as the cost impact of an implementation effort. Self-report of costs group program and workshop.
Falls Behaviour of the older person | Baseline and after 6 months
  Falls Behavioural Scale for the Older Person (FaB). The FaB scale consists of 30 items. Ten behavioral dimensions were identified including Cognitive Adaptations, Protective Mobility, Avoidance, Awareness, Pace, Practical Strategies, Displacing Activities, Being Observant, Changes in Level, and Getting to the Phone. Respondents are asked to rate 30 behavioral factors related to the prevention of falling on a 4-point rating scale (1-4) with 0 for does not apply. High scores equal the safest behaviours and low scores the riskiest behaviours (min. 0 - max: 120).
  The total FaB mean scores for items at baseline will be compared to the FaB mean score for items after 6 months.
Experiences with the BE-EMPOWERed program | The last 6 months of the study.
  Focus group and interviews with older people, healthcare professionals, policy makers
Feasibility of the BE-EMPOWERed program by experiences of the participants | The last 6 months of the study.
  Is defined as the extent to which a new treatment, or an innovation, can be successfully used or carried out within a given agency or setting.
  Focus group and interviews with older people, healthcare professionals, policy makers. A topic guide and interview guide will be used to guide the interviews and focus groups. The feasbility of the program will be questioned.
Acceptability of the BE-EMPOWERed program by experiences of the participants | The last 6 months of the study.
  Is the perception among implementation stakeholders that a given treatment, service, practice, or innovation is agreeable, palatable, or satisfactory.
  Focus group and interviews with older people, healthcare professionals, policy makers.
  Focus group and interviews with older people, healthcare professionals, policy makers. A topic guide and interview guide will be used to guide the interviews and focus groups. The acceptability of the program will be questioned.
Concerns about falling | Baseline and after 6 months
  Falls Efficacy Scale International (16 items) older person (min. 16 - max. 64). Score 16-22: People no concern about falling. Score 23-64: People are severe concerned about falling.
Reach of healthcare professionals | Immediately after every workshop (up to 1 month).
  Reach is defined as the absolute number, proportion, and representativeness of individuals who are willing to participate in a given initiative, intervention, or program, and reasons why or why not.
  Reach of healthcare professionals. Participant list workshops by the trainer.
Physical activity | Baseline and after 6 months
  Incidental and planned activity questionnaire (IPEQ) for older people. The IPEQ is a self-reported questionnaire and consists of 10 questions on physical activity. It measures type and amount of physical activity.
  Provides estimates of the frequency and duration of planned exercise and more casual day-to-day activities Outcome: hours of planned exercise per week Total time spent will be summed across all components and expressed as hours per week. The score will be derived from multiplying frequency score and duration score to create a total duration for the week score.
  The total hours of planned exercise per week will be measured at baseline and compared to the total hours of planned exercise per week after 6 months.

CONTACTS AND LOCATIONS:
Locations (1):
- KU Leuven, Leuven, Vlaams Brabant, Belgium

IPD SHARING:
Plan to Share IPD: Yes
The datasets used and/or analysed during the current study are available from the corresponding author on reasonable request. As far as requests are in line with the scope and research objectives of the Be-Empowered study.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: On reasonable request
Access Criteria: The datasets used and/or analysed during the current study are available from the corresponding author on reasonable request. As far as requests are in line with the scope and research objectives of the Be-Empowered study.

REFERENCES:
- [Background] Vandervelde S, Vlaeyen E, de Casterle BD, Flamaing J, Valy S, Meurrens J, Poels J, Himpe M, Belaen G, Milisen K. Strategies to implement multifactorial falls prevention interventions in community-dwelling older persons: a systematic review. Implement Sci. 2023 Feb 6;18(1):4. doi: 10.1186/s13012-022-01257-w. PMID 36747293
- [Background] Hopewell S, Adedire O, Copsey BJ, Boniface GJ, Sherrington C, Clemson L, Close JC, Lamb SE. Multifactorial and multiple component interventions for preventing falls in older people living in the community. Cochrane Database Syst Rev. 2018 Jul 23;7(7):CD012221. doi: 10.1002/14651858.CD012221.pub2. PMID 30035305
- [Background] Hopewell S, Copsey B, Nicolson P, Adedire B, Boniface G, Lamb S. Multifactorial interventions for preventing falls in older people living in the community: a systematic review and meta-analysis of 41 trials and almost 20 000 participants. Br J Sports Med. 2020 Nov;54(22):1340-1350. doi: 10.1136/bjsports-2019-100732. Epub 2019 Aug 21. PMID 31434659
- [Background] Bhasin S, Gill TM, Reuben DB, Latham NK, Ganz DA, Greene EJ, Dziura J, Basaria S, Gurwitz JH, Dykes PC, McMahon S, Storer TW, Gazarian P, Miller ME, Travison TG, Esserman D, Carnie MB, Goehring L, Fagan M, Greenspan SL, Alexander N, Wiggins J, Ko F, Siu AL, Volpi E, Wu AW, Rich J, Waring SC, Wallace RB, Casteel C, Resnick NM, Magaziner J, Charpentier P, Lu C, Araujo K, Rajeevan H, Meng C, Allore H, Brawley BF, Eder R, McGloin JM, Skokos EA, Duncan PW, Baker D, Boult C, Correa-de-Araujo R, Peduzzi P; STRIDE Trial Investigators. A Randomized Trial of a Multifactorial Strategy to Prevent Serious Fall Injuries. N Engl J Med. 2020 Jul 9;383(2):129-140. doi: 10.1056/NEJMoa2002183. PMID 32640131
- [Background] Lamb SE, Bruce J, Hossain A, Ji C, Longo R, Lall R, Bojke C, Hulme C, Withers E, Finnegan S, Sheridan R, Willett K, Underwood M; Prevention of Fall Injury Trial Study Group. Screening and Intervention to Prevent Falls and Fractures in Older People. N Engl J Med. 2020 Nov 5;383(19):1848-1859. doi: 10.1056/NEJMoa2001500. PMID 33211928
- [Background] Carpenter CR, Malone ML. Avoiding Therapeutic Nihilism from Complex Geriatric Intervention "Negative" Trials: STRIDE Lessons. J Am Geriatr Soc. 2020 Dec;68(12):2752-2756. doi: 10.1111/jgs.16887. Epub 2020 Oct 20. No abstract available. PMID 33079398
- [Background] Clemson L, Cumming RG, Kendig H, Swann M, Heard R, Taylor K. The effectiveness of a community-based program for reducing the incidence of falls in the elderly: a randomized trial. J Am Geriatr Soc. 2004 Sep;52(9):1487-94. doi: 10.1111/j.1532-5415.2004.52411.x. PMID 15341550
- [Background] Proctor E, Silmere H, Raghavan R, Hovmand P, Aarons G, Bunger A, Griffey R, Hensley M. Outcomes for implementation research: conceptual distinctions, measurement challenges, and research agenda. Adm Policy Ment Health. 2011 Mar;38(2):65-76. doi: 10.1007/s10488-010-0319-7. PMID 20957426
- [Background] Holtrop JS, Estabrooks PA, Gaglio B, Harden SM, Kessler RS, King DK, Kwan BM, Ory MG, Rabin BA, Shelton RC, Glasgow RE. Understanding and applying the RE-AIM framework: Clarifications and resources. J Clin Transl Sci. 2021 May 14;5(1):e126. doi: 10.1017/cts.2021.789. eCollection 2021. PMID 34367671
- [Background] Clemson L, Cumming RG, Heard R. The development of an assessment to evaluate behavioral factors associated with falling. Am J Occup Ther. 2003 Jul-Aug;57(4):380-8. doi: 10.5014/ajot.57.4.380. PMID 12911079
- [Background] Delbaere K, Hauer K, Lord SR. Evaluation of the incidental and planned activity questionnaire (IPEQ) for older people. Br J Sports Med. 2010 Nov;44(14):1029-34. doi: 10.1136/bjsm.2009.060350. Epub 2009 May 26. PMID 19474003
- [Background] Kempen GI, Todd CJ, Van Haastregt JC, Zijlstra GA, Beyer N, Freiberger E, Hauer KA, Piot-Ziegler C, Yardley L. Cross-cultural validation of the Falls Efficacy Scale International (FES-I) in older people: results from Germany, the Netherlands and the UK were satisfactory. Disabil Rehabil. 2007 Jan 30;29(2):155-62. doi: 10.1080/09638280600747637. PMID 17364765